CLINICAL TRIAL: NCT01071421
Title: Prevalence of Sleep Apnea-hypopnea Syndrome in Patients With Community Acquired Pneumonia, Prospective and Comparative Case-control Study
Brief Title: Sleep Apnea Syndrome and Community Acquired Pneumonia
Acronym: NEBULOSA
Status: Completed | Type: Observational
Sponsor: Hospital Universitario San Juan de Alicante (Other)
Responsible Party: Eusebi Chiner/ Pneumology Chairman Hospital Universitario San Juan de Alicante, Hospital Universitario San Juan de Alicante
Other Study IDs: NEBULOSA PROJECT
Record Dates: First submitted 2010-02-18; First posted 2010-02-19 (Estimated); Last update posted 2010-02-19 (Estimated); Status verified 2006-02

CONDITIONS: Sleep Apnea Syndrome; Polygraphy; Community Acquired Pneumonia; Infections
Keywords: Sleep apnea syndrome; community acquired pneumonia; prevalence
MeSH Terms: conditions — Sleep Apnea Syndromes; Community-Acquired Pneumonia; Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Control Group (B): Other Infections: Other infections admitted to the hospital
  Interventions: Device: abbreviated polysomnography
- Community Acquired Pneumonia (Group A): Patients admitted to hospital with Community Acquired Pneumonia defined by respiratory symptoms, fever and lung infiltrates
  Interventions: Device: abbreviated polysomnography

INTERVENTIONS:
Device: abbreviated polysomnography — Both groups will be studied with in-hospital respiratory polygraphy during the sleep. The group A will be studied with another respiratory polygraphy in the home one month after the resolution of CAP. Some questionnaires to measure the sleepiness (Epworth test), FOSQ test, in-home sleepiness questionnaire and symptoms questionary will be obtained in Group A and B
  Other Names: Respiratory Polygraphy; portable polysomnography

SUMMARY:
The association of sleep apnea-hypopnea syndrome (SAHS) with the infections of the lower airway has not been studied. The aspiration of secretions of the upper airway and the colonization by microorganisms is considered a main event in most of the cases of community acquired pneumonia (CAP) , and specially in the nosocomial pneumonia. The silent aspiration to the lower airway is a common phenomenon in normal subjects during the sleep and some studies has reported that the patients with SAHS present an increase of the risk to pharyngeal aspirations. In fact, the presence of nasal and bronchial inflammation in patients with SAHS is a recognized event. The patients with SAHS could have a risk increased to develop pneumonia due to predisposition to the pharyngeal microaspiration to lower airways during the sleep and other mechanical factors associated. The prevalence of SAHS in patients with CAP could be increased as regards the data published for the same Spanish population. The presence of an apnea-hypopnea index (AHI) could be a risk factor not only to to CAP but to to present a unfavorable clinical evolution in comparison to patients with CAP with a normal AHI. The aim of this study will establish a relation between SAHS and the pneumonia risk.

DETAILED DESCRIPTION:
This is a prospective comparative case control study to compare the prevalence of sleep apnea-hypopnea syndrome in patients with community acquired pneumonia (CAP).

Patients hospitalized with CAP (Group A)will be studied with respiratory polygraphy during the sleep and a second respiratory polygraphy will be conducted in home after the curation of the pneumonia (one month). During the admission, etiological study including blood cultures, serology, urinary antigens for legionella and S, pneumoniae, sputum cultures and other invasive techniques as bronchoscopy when appropriate will be obtained. Questionnaires related with sleep apnea-hypopnea syndrome will be obtained consisting in Epworth test, symptoms questionnaires and FOSQ test.

Group B are patients with other infections as urinary, bone, pelvic infections excluding upper or lower respiratory infections. Respiratory polygraphy will be performed in this group as in the group A obtaining the same questionnaires.

We compare the variables of respiratory polygraphy, questionnaires scores, percentage of patients with an AHI > 12 between both groups and we compare the variables obtained in the respiratory polygraphy performed in hospital and at home in the group A to evaluate if the condition of an altered AHI was previous to the CAP episode. We will obtain the prevalence of sleep apnea-hypopnea patients in both groups and we compare factor risks (COPD, diabetes mellitus, bronchial asthma, etc) between A and B. Finally multivariable analysis is conducted to evaluate the contribution of the AHI to CAP, as other recognize factor risk.

Both groups are paired by age, sex and body mass index

ELIGIBILITY:
Group A:

Inclusion Criteria:

* Hospital admission and Community acquired pneumonia

Exclusion Criteria:

* Nosocomial infections
* Low level of conscientiousness
* Neurological disease
* Impossibility to complete the questionnaires

Group B

Inclusion Criteria:

* Hospital admission and other infections different to respiratory infections

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to hospital with the diagnosis of community acquired pneumonia, excluding nosocomial pneumonia compared to patients with other infections excluding respiratory infections, admitted to hospital, paired by age, sex and body mass index
Sampling Method: Non-Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2006-04; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the prevalence of sleep anea-hypopnea syndrome in patients with community acquired pneumonia, defined by an apnea-hypopnea index more to 12 measured by respiratory polygraphy | 2 years

SECONDARY OUTCOMES:
To evaluate if the apnea-hypopnea index is a factor risk to community acquired pneumonia | 2 years
To evaluate if a high apnea-hypopnea index is observed in patients with community acquired pneumonia and if is maintained after the pneumonia resolution | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Eusebi Chiner, MD, Study Director — Head of Pneumology Section; Mónica Llombart, MD, Principal Investigator — Consultant
Locations (1):
- Sección de Neumología. Hospital Universitario San Juan de Alicante, Sant Joan d'Alacant, Alicante, Spain

REFERENCES:
- [Derived] Chiner E, Llombart M, Valls J, Pastor E, Sancho-Chust JN, Andreu AL, Sanchez-de-la-Torre M, Barbe F. Association between Obstructive Sleep Apnea and Community-Acquired Pneumonia. PLoS One. 2016 Apr 6;11(4):e0152749. doi: 10.1371/journal.pone.0152749. eCollection 2016. PMID 27050437